CLINICAL TRIAL: NCT00390728
Title: A Phase IIIb/IV, Multinational, Multicentre, Randomised, Open Study to Establish the Optimal Method for Initiating and Maintaining Lantus® (Insulin Glargine) Therapy Based on a Comparison of Two Treatment Algorithms to Determine Optimal Metabolic Outcomes, Safety, and Satisfaction in Subjects With Type 1 Diabetes Mellitus/ "HALT" Sub-study: Multicentre, Open Clinical Trial to Assess the Effect of Insulin Glargine on Symptomatic Hypoglycaemia, Fear of Hypoglycaemia and Quality of Life in Patients With Type 1 Diabetes
Brief Title: Insulin Glargine in Type I Diabetes Mellitus> Main Study "AT.LANTUS": A Trial Comparing Lantus Algorithms to Achieve Normal Blood Glucose Targets in Subjects With Uncontrolled Blood Sugar. Sub-study: "HALT"(Hypoglycaemia Avoidance With Lantus Trial)
Acronym: AT-LANTUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_3505
Record Dates: First submitted 2006-10-18; First posted 2006-10-20 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glargine

SUMMARY:
Primary objective:

AT.LANTUS main study*

* To determine the optimal treatment algorithm for insulin glargine based on the incidence of severe hypoglycaemia.(*Target Number of patients for the main study:2346)

HALT Sub-study**

* To test the hypothesis that titration regimens involving insulin glargine are associated with changes in the rate of symptomatic hypoglycaemic episodes together with changes in Fear of Hypoglycaemia as measured by the HFS-98 Questionnaire in Type I diabetes.(**Target Number of patients for the Sub-study: 250)

Secondary objectives:

AT.LANTUS main study

To determine:

* the incidence of symptomatic, asymptomatic and nocturnal hypoglycaemia with each treatment regimen
* the difference in glycemic control as measured by HbA1c and fasting blood glucose with each treatment regimen
* the difference in glycemic control as measured by HbA1c and fasting blood glucose between baseline and end of treatment
* the safety on the use of insulin glargine in each treatment algorithm
* the change in subject weight with each treatment regimen
* the change in insulin doses with each treatment regimen
* the change in Diabetes Treatment Satisfaction (Diabetes Treatment Satisfaction Questionnaire, sub-study only) with each treatment regimen

HALT Sub-study (baseline to study end)

* To estimate the relationship between change in HbA1c and incidence of hypoglycaemia
* To examine the effect of insulin glargine on Quality of Life (EQ-5D) in relation to incidence of hypoglycaemia
* To examine the effect of insulin glargine on the Hospital Anxiety and Depression Scale (HADS) in relation to the incidence of hypoglycaemia
* To examine the use of the Prescription Plan versus standard management (no Prescription Plan)

ELIGIBILITY:
Inclusion criteria:

* Subjects with type 1 diabetes mellitus who require a basal (long-acting) insulin for the control of hyperglycemia, with HbA1c values > 7.0% and < 12 %, and a body mass index (BMI) < 40 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2346
Dates: Start 2002-04; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Main study: Frequency of severe hypoglycaemia
Sub-study: The fear of hypoglycaemia as measured by the Hypoglycaemia Fear Survey questionnaire (HFS-98) assessed at baseline, 3 months and study end point or upon withdrawal of the subject from the study.

SECONDARY OUTCOMES:
Main study: HbA1c
Incidence of nocturnal, symptomatic and asymptomatic hypoglycaemia
Self monitored blood glucose
Change in subject weight
Changes in doses of insulin
Changes in treatment satisfaction
Safety assessment
Quality of Life (QoL)using the Diabetes Treatment Satisfaction Questionnaire (DTSQ)
Sub-study:Quality of Life tools assessed at baseline, 3 months and at study end point or upon withdrawal of the subject
Quality of Life - EQ-5D
Hospital Anxiety and Depression Scale (HADS)
Adverse events correlating with Quality of Life tools and hypoglycaemic events
Medications for diabetes
HbA1c
Weight and height (BMI)
Proportion of patients reaching HbA1c target as per participation with the Prescription Plan

CONTACTS AND LOCATIONS:
Overall Officials: Patrick SINNASSAMY, MD, Study Director — Sanofi